CLINICAL TRIAL: NCT01476865
Title: Articular Sonography: Findings in Healthy Subjects Compared With Rheumatoid Arthritis Patients
Brief Title: Articular Sonography: Healthy Subjects Versus Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, FLAVIA SOARES MACHADO, Flávia Soares Machado, Federal University of São Paulo
Other Study IDs: 1295/09
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Disorders of Synovium, Multiple Sites; Disorders of Subchondral Bone, Multiple Sites; Disorders of Cartilage, Hand Joints; Arthritis, Rheumatoid; Healthy People
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: normal, healthy people
- RA: rheumatoid arthritis patients

SUMMARY:
The purpose of this study is to establish the normality of sonographic synovial measures in joints more affected in rheumatoid arthritis patients and establish, in those joints, a sonographic value of synovium predictive of rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory, systemic and auto-imune disorder affecting primarily the joints. In RA, inflammatory synovium causes destruction of cartilage, erosion of the adjacent bone and ultimately loss of function of the affected joint. Newer imaging techniques, such as ultrasound (US), have shown promise in evaluation of RA. Many US scoring system have been used to classify and quantify the synovium, effusion, erosion and cartilage for assessing and monitoring AR. However, its use is considered problematical because there are very few data on normal joints and, at this point, there is no clear definition of excess amount of synovium in normal people.

ELIGIBILITY:
Inclusion Criteria:

* no articular disease (healthy group)
* establish rheumatoid arthritis (RA group)

Exclusion Criteria:

* diabetes
* hypothyroidism- hemophilia
* pregnancy
* previous septic arthritis
* previous articular surgery
* symptomatic osteoarthritis
* no superimposed collagenoses (RA group)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: terciary care clinic (rheumatoid arthritis patients) community sample (healthy people)
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, professor, Study Chair — Federal University of São Paulo; Rita NV Furtado, PhD, Study Chair — Federal University of São Paulo; Flávia S Machado, master, Principal Investigator — Federal University of São Paulo